CLINICAL TRIAL: NCT03048695
Title: Cognitive Remediation of Executive Dysfunction - Goal Management Training for Patients With Schizophrenia or High Risk for Schizophrenia
Brief Title: Goal Management Training for Patients With Schizophrenia or High Risk for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150601
Record Dates: First submitted 2017-01-16; First posted 2017-02-09 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Neurocognitive Disorders
MeSH Terms: conditions — Schizophrenia; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal Management Training (Experimental): Cognitive rehabilitation
  Interventions: Behavioral: GMT
- Waiting list (No Intervention)

INTERVENTIONS:
Behavioral: GMT — Metacognitive strategy training where the primary objective is to stop ongoing behavior to define goal hierarchies and monitor performance
  Arms: Goal Management Training

SUMMARY:
About 85% of patients with schizophrenia have cognitive impairments, executive functions being particularly affected. Executive dysfunction, and cognitive deficits in general, are important predictors of functional outcomes, including social problem solving, activities of daily living, life satisfaction, and the ability to return to work or school.The main objective of the current study is to examine the efficacy of group-based Goal Management Training (GMT) for patients with broad schizophrenia spectrum disorders or high risk individuals with executive deficits. The short term goals are to investigate whether GMT can improve participants' ability to organize and achieve goals in everyday life in addition to improving aspects of emotional health. A long-term goal would be to establish an evidence base for nonpharmacological interventions for patients with broad schizophrenia spectrum disorders or high risk for schizophrenia. Main research questions: (1) Does a RCT with GMT delivered to patients with broad schizophrenia spectrum disorders or high risk for schizophrenia result in improved executive functioning, measured by self-reported and/or objective measures of executive functions? (2) Does GMT result in improved goal attainment in everyday life, social- and real world functioning? (3) Does GMT have a positive impact on the patients' emotional health? (4) Are there specific characteristics in patients with broad schizophrenia spectrum disorders or high risk for schizophrenia that are associated with better treatment benefit from GMT?

ELIGIBILITY:
Inclusion Criteria:

* Being consecutively referred to treatment for a DSM-IV diagnosis of broad schizophrenia spectrum psychosis (schizophrenia, schizophreniform disorder and schizoaffective disorder) or high risk for psychosis or being treated for psychotic disorder for less than 5 years.
* Reporting executive problems through (a) structured interview, or (b) self-report, i.e. BRIEF scale T-score < 55.

Exclusion Criteria:

* Reported ongoing alcohol or substance abuse.
* Premorbid neurological disease or insult and/or comorbid neurological disease. ° Severe cognitive problems interfering with the capacity to participate.
* IQ below 70.

Ages: 16 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Behavior Rating Inventory for Executive Functions | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Conners Continuous Performance Test III | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Positive and Negative Syndrome Scale | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change

SECONDARY OUTCOMES:
Global Assessment of Functioning-Split Version | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
The Hotel Task | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Delis Kaplan Executive Function System (D-KEFS) subtests | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Digit span and Letter-number sequencing | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Iowa Gambling Task | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Dysexecutive Questionnaire (self-and informant) | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Cognitive Failures Questionnaire | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Goal Attainment Scaling | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Everyday Functioning from NORMENT Long time follow up questionnaires | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
General Perceived Self-Efficacy Scale | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Social Functioning Scale | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
The Perceived Quality of Life Scale | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Rosenberg self-esteem scale | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change
Hopkins Symptom Checklist 10 | Baseline, immediately post-intervention and 6 months follow-up
  Assessing change

CONTACTS AND LOCATIONS:
Overall Officials: Merete G Øie, Phd, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Sykehuset Innlandet Reinsvoll, Reinsvoll, Norway

REFERENCES:
- [Derived] Orm S, Oie MG, Haugen I. Iowa Gambling Task performance in individuals with schizophrenia: the role of general versus specific cognitive abilities. Front Psychiatry. 2024 Dec 10;15:1454276. doi: 10.3389/fpsyt.2024.1454276. eCollection 2024. PMID 39720440
- [Derived] Oie MB, Haugen I, Stubberud J, Oie MG. Effects of Goal Management Training on self-efficacy, self-esteem, and quality of life for persons with schizophrenia spectrum disorders. Front Psychol. 2024 Mar 7;15:1320986. doi: 10.3389/fpsyg.2024.1320986. eCollection 2024. PMID 38515967
- [Derived] Haugen I, Stubberud J, Haug E, McGurk SR, Hovik KT, Ueland T, Oie MG. A randomized controlled trial of Goal Management Training for executive functioning in schizophrenia spectrum disorders or psychosis risk syndromes. BMC Psychiatry. 2022 Aug 28;22(1):575. doi: 10.1186/s12888-022-04197-3. PMID 36031616